CLINICAL TRIAL: NCT05372120
Title: A Phase II Clinical Trial to Evaluate the Efficacy and Safety of ICP-192 in Treated Patients With Advanced Solid Tumors With FGF/FGFR Gene Alterations
Brief Title: A Clinical Trial of ICP-192 in Treated Patients With Advanced Solid Tumors With FGF/FGFR Gene Alterations
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICP-CL-00304
Record Dates: First submitted 2022-05-08; First posted 2022-05-12 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICP-192 (Experimental): 20 mg once daily
  Interventions: Drug: ICP-192

INTERVENTIONS:
Drug: ICP-192 — ICP-192 is a round, uncoated tablet, 4mg, 5mg. It is administered orally at the dose of 20 mg/day from day 1 to day 21 of each cycle until progression

SUMMARY:
This is a phase II clinical trial in treated patients with advanced solid tumors with FGF/FGFR gene alterations. The purpose of this study is to evaluate the efficacy and safety of ICP-192.

ELIGIBILITY:
Inclusion Criteria:

1. Signed the ICF and Age ≥ 18 years old, either sex.
2. ECOG ≤ 1.
3. Life expectancy of at least 3 months.
4. Part 1 (head and neck cancer cohort): Patients with HNC cancer who have failed or cannot tolerate standard therapy, and with FGF/FGFR gene alteration
5. Part 2 (other solid tumor cohorts): Patients with other solid tumor who have failed or cannot tolerate standard therapy, and with FGF/FGFR gene alteration
6. At least one measurable lesion as the target lesion at screening assessed according to RECIST V1.1 criteria.

Exclusion Criteria:

1. Prior treatment with selective FGFR inhibitors or FGFR antibodies.
2. Any corneal or retinal abnormalities that may result in an increased risk of ocular toxicity.
3. Previously or currently endocrine alterations affecting the regulation of calcium-phosphorus homeostasis. History and/or current evidence of extensive tissue calcification.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | From the time of first dose until objective disease progression, an average of 6 months
  ORR based on assessment of confirmed Complete response (CR) and partial response (PR) according to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST).

SECONDARY OUTCOMES:
Duration of response (DOR) | From the time of first dose until objective disease progression, an average of 6 months
  DOR is time interval from the first date that criteria for complete response or partial response are met to the first date of progression of disease
Disease Control Rate (DCR) | From the time of first dose until objective disease progression, an average of 6 months
  DCR based on assessment of confirmed Complete response (CR), partial response (PR) or stable disease(SD) according to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST).

OTHER OUTCOMES:
Progression Free Survival (PFS) | From the time of first dose until objective disease progression, an average of 6 months
  Progression free survival is the time period from start of study medication till the disease progression or death, whichever occurs first.
Overall survival (OS) | From the time of first dose until objective disease progression, an average of 1 year
  OS is the time period from start of study medication untill death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Ye Guo, Principal Investigator — Shanghai East Hospital
Locations (36):
- China (36):
  - The first affiliated hospital of bengbu medical college, Bengbu, Anhui
  - Anhui Provincal Cancer Hospital, Hefei, Anhui
  - Cancer Hospital.Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Lanzhou University, Lanzhou, Gansu
  - Affiliated Cancer Hospital and Institute of Guangzhou Medical University, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin Medical University cancer hospital, Harbin, Heilongjiang
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Henan Tumor Hospital, Zhengzhou, Henan
  - Union Hospital Toji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital Tongji Medical College of HUST, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Hunan Tumor Hospital, Changsha, Hunan
  - Nantong Cancer Hospital, Nantong, Jiangsu
  - Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu
  - The first hospital of jilin University, Changchun, Jilin
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Shandong Provincial Institute of Cancer Prevention and Treatment, Jinan, Shandong
  - QiLu Hospital of Shandong University, Jinan, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - Shanghai Ninth People's Hospital, Shanghai JiaoTong University School Medicine, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi An Jiaotong University, Xi’an, Shanxi
  - Sichuan Tumor Hospital, Chengdu, Sichuan
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Second People's Hospital of Yibin City, Yibin, Sichuan
  - Tianjin medical university cancer institute&hospital, Tianjin, Tianjin Municipality
  - Shaoyifu Hospital of Zhejiang University Medical College, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang